CLINICAL TRIAL: NCT02416349
Title: Acute Effects After Stretching Respiratory Muscles on Ventilatory Pattern and Volume Distribution of Chest Wall in Patients With Stroke: a Randomized Crossover Clinical Trial
Brief Title: Acute Effects After Stretching Respiratory Muscles on Ventilatory Pattern and Volume Distribution of Chest Wall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Catarina Souza Ferreira Rattes Lima, Msc, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STRETCHING RESPIRATORY MUSCLES
Record Dates: First submitted 2014-03-14; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Stroke
Keywords: Stroke; Stretching; Respiratory muscle; Ventilatory pattern; Optoelectronic plethysmography
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory Muscles Stretching (Active Comparator): Respiratory Muscles Stretching Neck stretching, upper chest stretching, pectoralis major stretching and lateral chest stretching.
  Interventions: Other: Respiratory Muscles Stretching
- Control Group (Placebo Comparator): All volunteers will be positioned at rest in a comfortable in a chair during 20 minutes.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Respiratory Muscles Stretching — Respiratory Muscles Stretching The stretching will occur throughout the expiratory phase to allow respiratory muscles to reach their maximal length, and two sets with 10 consecutive incursions will be use for each stretching pattern with an interval of 30 seconds between series.
  Pattern 1: Neck stretching Pattern 2: Upper chest stretching Pattern 3:Pectoralis major stretching Pattern 4:Lateral chest stretching
  Arms: Respiratory Muscles Stretching
Other: Control Group — Control Group - all volunteers will be positioned at rest in a comfortable in a chair during 20 minutes.
  Arms: Control Group

SUMMARY:
The purpose of study is to evaluate the acute effects of respiratory muscles stretching on ventilator pattern and volume distribution of chest wall in patients with right hemiparesis post-stroke and our hypothesis is that the use of RMS will be able to improve changes in the respiratory function.

DETAILED DESCRIPTION:
All study protocol will be performing in three different days. In the first day, the participants will undergo to the initial assessment, which consisted of anamnesis and anthropometric measurements: weight, height and body mass index (BMI). Then, they will be submitting to spirometry and respiratory muscle pressure using a manovacuometer.

All patients will submit underwent two types of intervention: respiratory muscles stretching (RMS) and remain at rest (control group). The stretching will occur throughout the expiratory phase to allow respiratory muscles to reach their maximal length, and two sets with 10 consecutive incursions will use for each stretching pattern with an interval of 30 seconds between series.

For the intervention in the control group, all volunteers will be position at rest in a comfortable in a chair during 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients post-stroke with right hemiparesis no more than 3 months, from both sexes, aged above 20 years, score between 1 and 3 according to Ashworth Scale for upper limbs, score above 85 according to Barthel Index and a minimum punctuation of 18 for Mini Mental State Examination.

Exclusion Criteria:

* Volunteers presenting facial paralysis; rheumatic or orthopedic diseases; spinal abnormalities or deformities that compromise the respiratory mechanics; spirometry with forced expired volume in the first second (FEV1) bellow 80% from predicted values and FEV1∕forced vital capacity (FVC) ≤ .7; presenting respiratory comorbidities; recent history of thoracic or abdominal surgery; hemodynamic instability or pregnancy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Chest Wall Volume | During assessment and intervention, on average for an hour
  Vcw -Total chest wall volume by Optoelectronic Plethysmography.
Compartmental chest wall volumes (composite) | During assessment and intervention, on average for an hour
  Vrcp - rib cage pulmonary volume; Vrca - rib cage abdominal volume; Vab - abdominal volume by Optoelectronic Plethysmography.

SECONDARY OUTCOMES:
Ventilatory Pattern (Composite) | During assessment and intervention, on average for an hour
  Total time (Ttot), inspiratory time (Tinsp), expiratory time (Texp), Tinsp/Ttot index, breathing rate (BR), minute volume (VE), mean inspiratory flow (MIF) and mean expiratory flow (MEF)
Lung Capacity (Composite) | During assessment and intervention, on average for an hour
  VC - Vital capacity; Inspiratory Capacity by Optoelectronic Plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Armele Andrade, PhD, Study Director — Federal University of Pernambuco - Department of Physical Therapy
Locations (1):
- Universidade Federal de Pernambuco - Laboratório de Fisiologia e Fisioterapia Cardiopulmonar - Recife - Brasil, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Rattes C, Campos SL, Morais C, Goncalves T, Sayao LB, Galindo-Filho VC, Parreira V, Aliverti A, Dornelas de Andrade A. Respiratory muscles stretching acutely increases expansion in hemiparetic chest wall. Respir Physiol Neurobiol. 2018 Aug;254:16-22. doi: 10.1016/j.resp.2018.03.015. Epub 2018 Mar 30. PMID 29608976